CLINICAL TRIAL: NCT01656460
Title: Stereotactic Body Radiation for Consolidation After Standard Chemoradiation for Stage 3 Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Thomas DiPetrillo (Other)
Collaborators: Memorial Hospital of Rhode Island (Other)
Responsible Party: Sponsor-Investigator, Dr Thomas DiPetrillo, Prinicipal Investigator, Brown University
Organization: Brown University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 259
Record Dates: First submitted 2012-07-24; First posted 2012-08-03 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stereotactic radiation Arm 1 (Experimental): Dose Levels/total Dose
  1 16 Gy
  Interventions: Radiation: Stereotactic radiation Arm 1
- Stereotactic radiation Arm 2 (Experimental): 2 20 Gy
  Interventions: Radiation: Stereotactic radiation Arm 2
- Stereotactic radiation Arm 3 (Experimental): 3 24 Gy
  Interventions: Radiation: Stereotactic radiation Arm 3
- Stereotactic radiation Arm 4 (Experimental): 4 28 Gy
  Interventions: Radiation: Stereotactic radiation Arm 4

INTERVENTIONS:
Radiation: Stereotactic radiation Arm 1 — Dose Levels Dose per Fraction Total Dose
  1 8 Gy 16 Gy
  Arms: Stereotactic radiation Arm 1
Radiation: Stereotactic radiation Arm 2 — Dose Levels Dose per Fraction Total Dose 2 10 Gy 20 Gy
  Arms: Stereotactic radiation Arm 2
Radiation: Stereotactic radiation Arm 3 — Dose Levels Dose per Fraction Total Dose 3 12 Gy 24 Gy
  Arms: Stereotactic radiation Arm 3
Radiation: Stereotactic radiation Arm 4 — Dose Levels Dose per Fraction Total Dose 4 14 Gy 28 Gy
  Arms: Stereotactic radiation Arm 4

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity stereotactic body radiation (SBRT) as consolidation following standard chemoradiation for patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
This protocol will investigate the potential role of SBRT for patients with stage 3 NSCLC. Eligible patients will first have received standard 50.4 Gy chemoradiation. Patients entering the study will have the opportunity to receive SBRT as a noninvasive option as compared to surgical resection. For patients who are not surgical candidates, SBRT after 50.4 Gy chemoradiation represents a technique of radiation consolidation that may be more effective and less toxic than standard conventional fractionated radiation

ELIGIBILITY:
PATIENT ELIGIBILITY Conditions for Patient Eligibility (Inclusion)

* Pathologically or cytologically confirmed NSCLC
* Stage III NSCLC according to the AJCC 7th edition staging criteria. Stage II (T1-3N1) patient that are deemed medically inoperable are also eligible.
* Concurrent chemoradiation to a radiation dose of 50.4 Gy.
* residual tumor volume after concurrent chemoradiation that is appropriate for SBRT:

  * Primary tumor <120cc (approximately 6cm diameter).
  * Mediastinal/Hilar disease: 1-2 involved regions <60cc (approximately 5cmx3cmx3cm)
* Absolute neutrophil count ≥ 1,000/uL, platelet ≥ 60,000/uL.
* Total bilirubin ≤ 2x upper institutional limit of normal (ULN), and AST or ALT ≤5x ULN.
* ECOG performance status 0 to 2
* Minimum life expectancy of 12 weeks.
* Age older than 18 years.
* Voluntary, signed written informed consent.
* Women of childbearing potential must have a negative pregnancy test
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 1 months thereafter.

Conditions for Patient Ineligibility (Exclusion)

* Disease progression during or after standard chemoradiation to 50.4 Gy
* Prior thoracic radiation other than the pre-operative radiation not greater than 50.4
* Metastatic disease
* Uncontrolled severe, intercurrent illness.
* Women who are breast-feeding.
* No chemotherapy within 2 weeks from the first SBRT treatment.
* Concurrent anticancer therapy.
* Prior complete resection of all NSCLC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2017-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG Study Chair
Locations (2):
- United States (2):
  - memorial Hospital of Rhode island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stereotactic Radiation Dose Level 1: Radiation: Stereotactic radiation Arm 1 Dose Levels Dose per Fraction Total Dose
  1 8 Gy 16 Gy
- Stereotactic Radiation Dose Level 2: Radiation: Stereotactic radiation Arm 2 Dose Levels Dose per Fraction Total Dose 2 10 Gy 20 Gy
- Stereotactic Radiation Dose Level 3: Radiation: Stereotactic radiation Arm 3 Dose Levels Dose per Fraction Total Dose 3 12 Gy 24 Gy
- Stereotactic Radiation Dose Level 4: Radiation: Stereotactic radiation Arm 4 Dose Levels Dose per Fraction Total Dose 4 14 Gy 28 Gy
Period: Overall Study
Arm/Group | Stereotactic Radiation Dose Level 1 | Stereotactic Radiation Dose Level 2 | Stereotactic Radiation Dose Level 3 | Stereotactic Radiation Dose Level 4
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stereotactic Radiation: stereotactic
Arm/Group | Stereotactic Radiation
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 63.9 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Early and Intermediate Toxicity for Dose Limiting Toxicity
Description: Any toxicity related to the radiation treatment will be scored and graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Serious adverse events will be captured from the time the patient signs consent until 12 weeks after the last SBRT.
  DLTS: defined in protocol as: Dose limiting toxicities will be defined as grade 3 or greater treatment related pneumonitis, cardiac toxicity, bronchial injury or chest wall pain during or within 4 weeks of completion of SBRT.
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Arm 1-Stereotactic Radiation Dose Level 1: Radiation: Stereotactic radiation Arm 1 Dose Levels Dose per Fraction Total Dose
  1 8 Gy 16 Gy
- Arm 2-Stereotactic Radiation Dose Level 2: Radiation: Stereotactic radiation Arm 2 Dose Levels Dose per Fraction Total Dose 2 10 Gy 20 Gy
- Arm 3-Stereotactic Radiation Dose Level 3: Radiation: Stereotactic radiation Arm 3 Dose Levels Dose per Fraction Total Dose 3 12 Gy 24 Gy
- Arm 4-Stereotactic Radiation Dose Level 4: Radiation: Stereotactic radiation Arm 4 Dose Levels Dose per Fraction Total Dose 4 14 Gy 28 Gy
Arm/Group | Arm 1-Stereotactic Radiation Dose Level 1 | Arm 2-Stereotactic Radiation Dose Level 2 | Arm 3-Stereotactic Radiation Dose Level 3 | Arm 4-Stereotactic Radiation Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline, 30 days post last dose of SBRT, 12 weeks post last dose of SBRT
Arm/Group | Arm 1-Stereotactic Radiation Dose Level 1 | Arm 2-Stereotactic Radiation Dose Level 2 | Arm 3-Stereotactic Radiation Dose Level 3 | Arm 4-Stereotactic Radiation Dose Level 4
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Stereotactic Radiation Dose Level 1 (N=3) | Arm 2-Stereotactic Radiation Dose Level 2 (N=3) | Arm 3-Stereotactic Radiation Dose Level 3 (N=3) | Arm 4-Stereotactic Radiation Dose Level 4 (N=3)
K(3), AKI secondary to cisplatin nephrotoxicity(5) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — not related to study
AKI(2*) RT poor intake, CR(2*) RT poor intake, Fatigue (2*) RT pneumonia or chemo, H/A(2*) related (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypoglycemia(2*), chest pain (3*), Hyperglycemia(3*), HGB(2*), CR(1*) k(1*) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — ALL events unrelated to SBRT and related to patients underlying medical history
Dyspnea 4*, Tachycardia 2*, Fever 1*cough 1*- (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — all unlikely related to SBRT
Bronchopulmonary Hemorrhage (5) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — likely related to SBRT as late toxicity
upper respiratory infection (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — NOT r/t SBRT.Pt #13: fever(3),AKI(1),dyspnea(3),URI(3),Lung Infection Influenza A(3), Productive cough(1) F/u: MG(3),PLT(1),AKI(1),CR(1),nausea(1),dizziness(1), leukocytosis(3),hypoxia, URI (3) F/U #2 pneumonia(3*)&influzena (3*)
URI (3*) rt chemo, PLT(2*) PR chemo, hyponatremia (3*) PR chemo, bilateral thigh pain(2*) suspected (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1-Stereotactic Radiation Dose Level 1 (N=3) | Arm 2-Stereotactic Radiation Dose Level 2 (N=3) | Arm 3-Stereotactic Radiation Dose Level 3 (N=3) | Arm 4-Stereotactic Radiation Dose Level 4 (N=3)
HgB (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
vomiting (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WBC (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
dermatitis (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
pleural effusion (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymph (Investigations) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Bili (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dyspnea/hypoxia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
myalgia (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
esophagitis (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
K (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
ANC (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
cough (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
fatigue (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
pain- thigh/leg/groin/chest wall (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
nausea (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ca (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pneumonitis ,upper respiratory infection (URI),lung Infection (influenza A) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
AST (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Magnesium (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fever (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diarrhea (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
chills (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
edema (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
aspiration (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No